CLINICAL TRIAL: NCT06751212
Title: Observation on the Efficacy of Radiofrequency Ablation for Patients With Moderate to Severe Gastric Atrophy With Enterosis With or Without Atrophy of Intraepithelial Neoplasia: An Observational Study
Status: Not yet recruiting | Type: Observational
Sponsor: Xiuli Zuo (Other)
Responsible Party: Sponsor-Investigator, Xiuli Zuo, chief physician, Shandong University
Organization: Shandong University (Other)
Other Study IDs: KYLL-202408-006-1
Record Dates: First submitted 2024-12-17; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Atrophic Gastritis
MeSH Terms: conditions — Gastritis, Atrophic | interventions — Radiofrequency Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No

INTERVENTIONS:
Procedure: Radiofrequency ablation alone — Endoscopic radiofrequency ablation (RFA) consists of delivering a 465 KHz energy waveform to the diseased tissue through an array of bipolar electrodes. The electrodes are mounted externally to the balloon, on an articulating platform attached to the distal end of the endoscope, or on a flexible catheter that penetrates the scope. The principle of radiofrequency ablation is that the action of high-frequency alternating current (HFAC) induces the movement of charged particles within the tissue to generate heat, which results in evaporation of water inside and outside the cell, drying, and solidifying and shedding to the point of aseptic necrosis.RFA has been demonstrated to safely, effectively, and durably eradicate early stage tumors of Barrett's esophagus as well as gastric low-grade endoepithelial neoplasia, and is said by a consensus of experts to be capable of treating moderately severe atrophic enterocolitis that has not yet progressed to gastric low-grade intraepithelial neoplasi

SUMMARY:
The aim of this observational study was to understand the effect of radiofrequency ablation on subjects with moderate to severe gastric atrophy with enterocolitis with or without low-grade intraepithelial neoplasia who underwent radiofrequency ablation. The main question it aims to answer is:

Does radiofrequency ablation therapy reduce gastric mucosal atrophy and enterosis in subjects with moderate to severe gastric atrophy with enterosis with or without low-grade intraepithelial neoplasia?

DETAILED DESCRIPTION:
Outpatient or inpatient collection of study participants was done by recruiting participants who met the inclusion criteria and did not meet the exclusion criteria and signed an informed consent form. Study participants were identified for enrollment and a case report form was completed. The basic demographic information of the study participants was recorded, along with the results of existing routine laboratory tests, and symptom-related clinical characteristics. Gastroenterology reports and pathology reports were retained for enrolled study participants to score and grade each study participant specifically, and all study participants were treated with radiofrequency ablation after enrollment. Follow-up gastroscopy was performed on study participants 3 months after treatment, adverse reactions during the two gastroscopies were recorded and case report forms were supplemented, gastroscopy reports and pathology reports of study participants were retained again, and gastroscopy reports and pathology reports of study participants were evaluated, and data on changes were summarized. Follow-up gastroscopy was performed on study participants 3 months after treatment, adverse reactions during the two gastroscopies of study participants were recorded and additional case report forms were completed, gastroscopy reports and pathology reports of study participants were again retained and gastroscopy reports and pathology reports of study participants were evaluated, and data on changes were summarized. Study participants who failed treatment but did not develop new intraepithelial neoplasia summarized the reasons for their failure and were re-treated with radiofrequency ablation 3 months later, and this was repeated until treatment was successful; study participants who developed new low-grade intraepithelial neoplasia were treated with radiofrequency ablation at post-treatment follow-up, and this was repeated until treatment was successful; and study participants who developed new intermediate- and high-grade intraepithelial neoplasia were treated with ESD at post-treatment follow-up, and this was repeated until treatment was successful. All data were summarized at the end of enrollment for all study participants and statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years old, male or female.
* Patients who had undergone gastroscopy within 3 months prior to inclusion, and whose histologic diagnosis of chronic gastritis was histologically atrophic enterocolitis graded at moderate-to-severe with or without low-grade intraepithelial neoplasia.
* Patients who had undergone gastroscopy within 3 months prior to inclusion, and whose OLGA (atrophic grading and staging criteria for chronic gastritis) or OLGIM (enteric grading and staging criteria for chronic gastritis) staging criteria had reached moderately severe.
* Helicobacter pylori negative.

Exclusion Criteria:

* Pregnant or lactating women.
* Previous history of malignant tumors of the digestive tract or history of gastrointestinal surgery.
* Malignant tumors of other organs, coagulation disorders, cardiopulmonary insufficiency, hepatic and renal insufficiency, etc.
* Those who are unable or unwilling to sign the informed consent form.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study recruited study participants with moderate-to-severe gastric atrophy with enterocolitis with or without low-grade intraepithelial neoplasia detected in the outpatient or inpatient setting; upon entry into the study, study participants were required to meet the inclusion criteria and not to meet the exclusion criteria, and to sign an informed consent form
Sampling Method: Non-Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2024-12-31 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
Eradication and remission rates after radiofrequency ablation therapy in study participants with moderate to severe gastric atrophic enterosis with or without low-grade intraepithelial neoplasia | 3 Months After Participants Underwent Radiofrequency Ablation

SECONDARY OUTCOMES:
Procedure time for radiofrequency ablation therapy in study participants with moderate to severe gastric atrophic enterocolitis with or without low-grade intraepithelial neoplasia | Within 24 hours after the participant underwent radiofrequency ablation
Length of hospitalization for radiofrequency ablation in study participants with moderate to severe gastric atrophic enterocolitis with or without low-grade intraepithelial neoplasia | Within 24 hours after participants were successfully discharged from the hospital after undergoing radiofrequency ablation procedures
Incidence of adverse reactions to radiofrequency ablation therapy in study participants with moderate to severe gastric atrophic enterocolitis with or without low-grade intraepithelial neoplasia | 3 Months After Participants Underwent Radiofrequency Ablation.

IPD SHARING:
Plan to Share IPD: Undecided